CLINICAL TRIAL: NCT03645642
Title: To Study the Safety and Efficacy of Midodrine With Albumin Versus Albumin Alone in Hepatic Hydrothorax- A Pilot Randomised Controlled Trial
Brief Title: To Study the Safety and Efficacy of Midodrine With Albumin Versus Albumin Alone in Hepatic Hydrothorax
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-18
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2019-11

CONDITIONS: Hepatic Hydrothorax
MeSH Terms: interventions — Midodrine; Albumins; Diuretics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midodrine (Experimental): Midodrine (5 mg TDS) along with albumin(20g/l) and diuretics. The dose of Midodrine will titrated according to the Mean arterial pressure (75-90mmhg). The dose will be increased to a maximum of 12.5 mg thrice daily.
  Interventions: Drug: Midodrine; Biological: Albumin; Drug: Diuretics
- Albumin with diuretics (Active Comparator): Albumin(20g/l) and diuretics.
  Interventions: Biological: Albumin; Drug: Diuretics

INTERVENTIONS:
Drug: Midodrine — Midodrine 5 mg thrice daily
  Arms: Midodrine
Biological: Albumin — Albumin 20g/l
Drug: Diuretics — Diuretics will be continued with an maximum dose of furosemide (160mg) and Aldactone 400 mg.

SUMMARY:
Hepatic hydrothorax is defined with accumulation of transudate fluid (500 ml) in the pleural cavity in patients with decompensated liver cirrhosis but without cardiopulmonary and pleural diseases. The Prevalence is 5-12% The treatment for hydrothorax is diuretics, repeated thoracocentensis, TIPS and liver transplant.. Midodrine increases effective arterial blood volume and also increases renal perfusion.It has also been used in Refractory ascitis .It has been shown to mobilise ascitis. In patients who are ineligible for TIPS and Liver transplant there is no data on Midodrine and its effects on Hydrothorax in cirrhotics.There are also no guidelines on the use of albumin during Pleural fluid tapping and the dose to be used. This study is being done to assess the safety and efficacy of Midodrine in hydrothorax.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hepatic hydrothorax
* Patients with age from 18-75 years
* No evidence of Cardiac and pulmonary disease

Exclusion Criteria:

* Renal failure ( Creatinine>2.5mg/dl)
* Gastrointestinal bleeding
* Spontaneous bacterial empyema/ Peritonitis
* Patients with urinary retention
* Intrinsic advanced pulmonary disease (CXR, HRCT thorax)
* Cardiovascular disease (Electrocardiogram, 2D Echo)
* Systemic arterial hypertension
* Presence of hepatocellular carcinoma or portal vein thrombosis, Budd chiari syndrome
* Patients with active untreated sepsis
* Pregnancy
* Patients with hepatic encephalopathy
* Patients eligible for TIPS
* No use of drugs affecting systemic hemodynamics prior to 7 day of enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in frequency of thoracentesis. | 3 months

SECONDARY OUTCOMES:
Partial or complete resolution of hepatic hydrothorax | 3 months
Development of Spontaneous Bacterial Empyema | 3 Months
Development of Thorocacocentesis Induced circulatory dysfunction | 3 Months
Drug related adverse events in both arms | 3 Months
Transplant free survival in both groups | 3 Months
Predictors and mechanisms of repeated development of hepatic hydrothorax | 3 Months
Number of patients going for TIPS(Transintrahepatic Portosystemic Shunts) | 3 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided